CLINICAL TRIAL: NCT01196325
Title: Anterior and Posterior Segment Vascular Changes Following Laser and Anti-Vascular Endothelial Growth Factor (VEGF) Treatment of Diabetic Retinopathy.
Acronym: VEGF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Toronto (Other)
Collaborators: Ontario Research Fund (Other)
Responsible Party: Principal Investigator, Chris Hudson, Professor, University of Toronto
Other Study IDs: 09-0258-BE
Record Dates: First submitted 2010-09-03; First posted 2010-09-08 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetes; Diabetic Macular Edema; Laser; Anti-VEGF; Morphology; Blood Flow; Vision
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Laser Group: Patients who are clinically indicated for the laser treatment
- Anti-VEGF Group (Bevacizumab): Patients who are clinically indicated for the intravitreal injection of Bevacizumab
- Anti-VEGF Group (Ranibizumab): Patients who are clinically indicated for intravitreal injection of Ranibizumab
- Age-matched controls: Group of non-diabetic participants who will be age and gender matched

SUMMARY:
The study will investigate changes in the structure and function of blood vessels in the front and back of the eye following laser and anti-VEGF treatments for sight-threatening diabetic eye disease. Sixty four volunteers will be recruited, including age-matched control subjects and diabetic patients who require conventional or contemporary treatment for pre-existing diabetic eye disease. Volunteers will be assessed before and after treatment using state-of-the-art techniques to measure vision, the rate of blood flow and structure at the front and back of the eye and the effectiveness of blood flow delivery. Changes following treatment in these novel, non-invasive techniques will be quantified and described. We anticipate that conventional and new / developing treatments will lead to narrowing of the vessels and consequent reduction of blood flow at the back and front of the eye. There will be a strong relationship between structural changes of the eye and functional changes of blood vessels at the front and back of the eye. The results of this study will improve our understanding of the impact of the various treatments on the entire eye. The research will also ensure an improved understanding of the mechanisms of action of the various treatments and will provide insight of reasons for good or poor outcomes, based upon specific changes in structure and blood flow.

DETAILED DESCRIPTION:
Diabetic Retinopathy (DR) is the single leading cause of blindness in people of working age. The total number of people living with diabetes in Canada is well over 2 million. The WHO estimates that around 12% of people with diabetes are blind or will develop severe vision loss. The two most common treatments of DR are: Laser Photocoagulation and anti-VEGF intravitreal injection. Clinical evidence demonstrates that these treatments lead to morphological and vascular retinal changes, however the actual mechanism and nature of post treatment changes is not fully understood. It is only recently that objective and quantitative imaging and hemodynamic technologies with previously unachievable resolution have become available that enable us to evaluate and to compare various effects of these treatments on vital eye structures.

We are proposing to take advantage of these state-of-the-art technologies in order to explore unknown effects of treatments on vital eye structures. We hypothesize that: 1) Laser Photocoagulation and anti-VEGF treatments will result in vessel constriction and hence reduction in posterior (retinal and choroidal) and anterior (conjunctival) ocular blood flow; 2) Changes in anterior segment ocular morphology and blood flow will positively correlate with changes in posterior segment morphology and blood flow; 3) Combined treatments will result in a greater reduction in posterior and anterior blood flow than any single treatment; 4) There will be differences in anterior and posterior blood flow outcomes and in anterior segment oxygen saturation when compared to healthy controls.

The study will include four groups of participants: Laser treatment group; Intravitreal injection of Bevacizumab treatment group; Intravitreal injection of Ranibizumab treatment group; Healthy age matched controls. The administration of ranibizumab and bevacizumab will be randomized across participants. Randomization number will be assigned to each participant and recorded in a Master Randomization Assignment List. All patients will be recruited from the Retina Clinics of the Toronto Western Hospital.

Every type 2 diabetic patient with Diabetic Macular Edema will be assessed prior to treatment and followed-up on the 3rd, 7th,30th day and 3 months after the initial treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age range of 35-75 yrs
* Type 2 diabetes apart from age-matched control group
* Visual acuity of 20/400 or better
* Confirmed diagnose of Clinical Significant Diabetic Macular Edema (applies for Diabetic Groups only)
* Previously untreated eye for retinal diseases and disorders

Exclusion Criteria:

* Distance refractive error > ± 6.00 DS & / or ± 2.50 DC
* Intraocular pressure ≥ 22mm Hg
* Proliferative Diabetic Retinopathy
* Any other active eye disease and disorder
* Participants with history of cardiovascular events, stroke, thromboembolic events, transient ischemic attack, uncontrolled hypertension.
* Any active ocular infection;
* History of glaucoma;
* Known allergy, hypersensitivity or contraindication to the study medication;
* Pregnancy, breast feeding, or women of childbearing potential who are not using a reliable method of contraception;
* Proteinuria and/or renal impairment;
* Surgery within the past 28 days.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetic patients with clinically sight-threatening Diabetic Macular Edema will be recruited from the Retina Clinics of Toronto Western Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2009-07; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Quantitative inner retinal blood flow | Baseline, 3, 7, 30 days and 3 months
  Inner retinal blood flow will be measured using Canon Laser Blood Flowmeter

SECONDARY OUTCOMES:
Mean retinal thickness for an annulus centered on fovea | Baseline,3,7,30 days, and 3 months
  Mean retinal thickness will be measured using Heidelberg Spectralis Spectral Domain Optical Coherence Tomography
Best Corrected Visual Acuity (LogMAR, EDTRS) | Baseline, 3, 7, 30 days and 3 months
  Best Corrected Visual Acuity will be examined using 96% and 10 % contrast EDTRS letter charts.
Quantitative anterior blood flow | Baseline, 3, 7, 30 days and 3 months
  Quantitative anterior blood flow will be assessed by measuring velocity of individual rbc's (μm/sec) and blood oxygen saturation(%)
Mean angle opening distance and trabecular-iris spur area | Baseline, 3, 7, 30 days and 3 months
  Mean angle opening distance and trabecular-iris spur area will be measured by Heidelberg Slit-Lamp Optical Coherence Tomography.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Hudson, PhD, Principal Investigator — University of Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada